CLINICAL TRIAL: NCT05734014
Title: Strengthening Healthy Relationships Among Apsaalooke Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4W8808
Record Dates: First submitted 2022-09-30; First posted 2023-02-17 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Youth Engagement

STUDY DESIGN:
Intervention Model Description: The feasibility study includes pilot testing activities and an evaluation of the activities. This study focused on developing the lessons that would promote cultural connectedness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Youth Sessions focused on respect, communication, and relationally.
  Interventions: Behavioral: Connectedness Activities

INTERVENTIONS:
Behavioral: Connectedness Activities — Indigenous Connectedness: Promoting respect, listening to elders, understanding Crow cultural values.

SUMMARY:
This pilot project uses community based participatory research principles to build upon cultural strengths to develop a feasibility of intervention to promote relationality and connectedness among Apsáalooke youth. This project worked closely with a Community Advisory Board (CAB) members to develop all stages of the project. The CAB identified 5th grade as an important age to focus. The feasibility study is developing pilot activities related to respecting promoting intergenerational, family, community and land connectedness among Crow youth.

DETAILED DESCRIPTION:
Study Purpose: The purpose of this study is to conduct a feasibility and acceptability of a pilot intervention to promote relationality among Apsáalooke youth. This formative study is grounded in community-based participatory efforts to build locally relevant educational programming for youth and support the development of future evidence-based programming for youth.

Participants and Inclusion Citeria:

Participants in this study consisted youth who are a maximum of 13 years old who are enrolled in 5th-6th grade at the time of the study. Eligibility criteria included youth that live on or near the Crow Reservation in Montana and have parental or guardian consent to participate. Recruitment efforts were conducted in partnership with local schools, educational liaisons, and community champions. Information about the program was shared through school announcements, flyers sent home with students and presentations during school-based and community events. Interested families received informational packets and consent forums outlining the purpose, procedures and voluntary nature of participants. Informed consent was also obtained from parents and assent from each youth participant. The recruitment spanned from May 2024 through June 2024. A total of 10 participants were recruited and enrolled in the study.

Data Collection Methods

Data for this feasibility study consisted of process evaluation data and qualitative, art-based reflections. The primary data collected included recruitment and retention metrics: Researchers tracked the number of students recruited, consented, and retained during the program. Session Observations: Trained facilitators and researchers documented implementation fidelity, student engagement, and logistical issues during sessions. Observational field notes were compiled systematically and informed the overall assessment of feasibility.

Arts-based qualitative reflections. At the conclusion of each session, students participated in a reflective activity using paper and markers to draw or write about their experiences. Prompts included: "What did you like best today?" "What did you learn?" "What would you like to share with your family?" The creative responses provided insight into the youth's internalization of key messages and their personal engagement with the content. Following the acidity, students voluntarily shared their drawing and narratives with the group. Researchers took detailed notes during these sharing moments to record accurate explanations.

ELIGIBILITY:
Inclusion Criteria: Students who are entering the fifth and sixth grade and who live on or near the Crow reservation will be invited to participate in the summer camp.

Exlcusion Criteria: Youth not enrolled in fifth or sixth grade, and who did not obtain parental or guardian consent.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Simonds, ScD, Principal Investigator — Montana State University
Locations (1):
- Vanessa Simonds, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5th and 6th grade Youth; recruited through flyers and social media
Groups:
- Intervention: Educational Intervention with session with focus on Respect, Communication and Relationally
Period: Overall Study
Arm/Group | Intervention
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Crow Knowledge
Description: Arts-based open-ended question for youth to describe what they liked, what was challenging or what they learned. We examined whether they mentioned the clan system (Crow Relationally), or the Creation Story.
Time Frame: 2 week
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 10
Participants
  Mentioned Crow Stories | 8
  Did not Mention Crow stories | 2
Statistical Analysis 1: Comparison: Intervention; Test type: Other; Qualitative Analysis of arts-based reflections. Thematic analysis and count of whether the participant drew or mentioned Crow stories related to relationality

ADVERSE EVENTS:
Time Frame: Through study completion, 2 weeks
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT05734014/Prot_SAP_000.pdf